CLINICAL TRIAL: NCT03208413
Title: The Effect of Thalidomide in Radiation-induced Brain Injury（RI）: a Phase II Clinical Trial
Brief Title: The Therapeutic Effect of Thalidomide in RI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017001
Record Dates: First submitted 2017-05-08; First posted 2017-07-05 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Radiation Injuries
Keywords: thalidomide; radiation-induced brain injury
MeSH Terms: conditions — Radiation Injuries | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thalidomide (Experimental): Thalidomide with a dosage of 25 mg at bedtime daily one week (days 1-7), then 50 mg at bedtime daily for one week (days 8-14), then 75 mg at bedtime daily for one week (days 15-21), then 100 mg at bedtime daily for 12 weeks (days 22-105), in the absence of unacceptable toxicity or severe deterioration.
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Thalidomide with a dosage of 25 mg at bedtime daily one week (days 1-7), then 50 mg at bedtime daily for one week (days 8-14), then 75 mg at bedtime daily for one week (days 15-21), then 100 mg at bedtime daily for 12 weeks (days 22-105), in the absence of unacceptable toxicity or severe deterioration.

SUMMARY:
Purpose: This phase II clinical trial aims to evaluate the indications, therapeutic effects and side effects of thalidomide in radiation-induced brain injury.

Further study details as provided by Sun Yat-sen Memorial Hospital, Sun Yat-sen University / Yameitang.

Primary outcome measure: The primary endpoint is the brain injury remission at week 15. In brief, the brain lesion will be evaluated by using brain MRI scan before and after thalidomide regimen. The clinical efficacy is defined as ≥ 25% reduction in brain edema volume on FLAIR images at week 15, as compared with that before thalidomide usage.

DETAILED DESCRIPTION:
There is no acknowledged and effective standard treatment for radiation-induced brain injury (RI). Glucocorticoids and bevacizumab during acute period are optional ways to reduce the brain edema. However, glucocorticoids and bevacizumab are unsuitable or ineffective for some patients, especially in the early stage of RI. The investigators supposed that angiogenesis might play a key role in the pathogenesis of RI, and that thalidomide, as an antiangiogenic drug, would reduce immature angiogenesis and improve vessel maturation in RI.

Primary objectives: This phase II clinical trial aims to evaluate the indications, therapeutic effects and safety of thalidomide in radiation-induced brain injury.

OUTLINE: This is a phase II, open-label, single arm clinical trial. Patients are enrolled and administrated with thalidomide. Thalidomide is supplied as 25 mg per pill to be taken by mouth.

Arm І: Patients receive thalidomide with a dosage of 25 mg at bedtime daily one week (days 1-7), then 50 mg at bedtime daily for one week (days 8-14), then 75 mg at bedtime daily for one week (days 15-21), then 100 mg at bedtime daily for 12 weeks (days 22-105), in the absence of unacceptable toxicity or severe deterioration.

ELIGIBILITY:
Inclusion Criteria

* Prior irradiation >/= 12 months prior to study entry.
* Radiographic evidence to support the diagnosis of radiation-induced brain injury without tumor recurrence.
* Age>/= 35 years.
* Contraindication to glucocorticoids and bevacizumab treatment due to history or high risk of severe adverse effects, or non-effective response to glucocorticoids and bevacizumab treatment in 12 months prior to study entry.
* Estimated life expectancy must be greater than 12 months.
* Routine laboratory studies: bilirubin </=1.0 * upper limits of normal (ULN); aspartate aminotransferase (AST or SGOT) or alanine aminotransferase (ALT)< 1.0 * ULN; creatinine <1.0 * ULN; white-cell count >/= 4,000 per cubic millimeter; neutrophils count >/=1500 per cubic millimeter platelets >/= 100,000 per cubic millimeter; Hb >/=110 gram per millilitres; PT, APTT, INR in a normal range.
* Ability to understand and willingness to sign a written informed consent document, or constant caregivers who well understand and willingness to sign a written informed consent document.

Exclusion Criteria

* Evidence of tumor metastasis, recurrence, or invasion;
* Current usage of bevacizumab;
* Current usage of glucocorticoids;
* Evidence of very high intracranial pressure that suggests brain hernia and need surgery;
* History of psychiatric diseases before radiotherapy;
* History of seizures;
* History of arteriosclerotic cardiovascular diseases (ASCVD), e.g. stroke, myocardial infaction, unstable angina, within 6 months;
* New York Heart Association Grade II or greater congestive heart failure;
* Serious and inadequately controlled cardiac arrhythmia;
* Significant vascular disease, e.g. moderate or severe carotid stenosis, aortic aneurysm, history of aortic dissection;
* Severe infection;
* History of allergy to relevant drugs;
* Pregnancy, lactation, or fertility program in the following 12 months;
* History or current diagnosis of peripheral nerve disease;
* Abnormal in liver and renal function;
* Active tuberculosis;
* Transplanted organs;
* Human immunodeficiency virus;
* Participation in other experimental studies.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
the brain injury remission | Week 15
  The brain injury remission is defined as ≥ 25% reduction in brain edema volume on FLAIR images at week 15, as compared with that before thalidomide usage

SECONDARY OUTCOMES:
improvement of quality of life | Week 15
  the difference value of WHO-QOL scale before and after thalidomide regimen
improvement of neurological function | Week 15
  the difference value of LENT/SOMA scales before and after thalidomide regimen

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, M.D., Ph.D., Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (3):
- China (3):
  - Cancer canter of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangzhou Huiai Hospital, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cheng J, Jiang J, He B, Lin WJ, Li Y, Duan J, Li H, Huang X, Cai J, Xie J, Zhang Z, Yang Y, Xu Y, Hu X, Wu M, Zhuo X, Liu Q, Shi Z, Yu P, Rong X, Ye X, Saw PE, Wu LJ, Simone CB 2nd, Chua MLK, Mai HQ, Tang Y. A phase 2 study of thalidomide for the treatment of radiation-induced blood-brain barrier injury. Sci Transl Med. 2023 Feb 22;15(684):eabm6543. doi: 10.1126/scitranslmed.abm6543. Epub 2023 Feb 22. PMID 36812346